CLINICAL TRIAL: NCT03411200
Title: Engaging the Older Cancer Patient; Patient Activation Through Counseling, Exercise and Mobilization - Pancreatic, Biliary Tract, and Lung Cancer (PACE-Mobil-PBL) - a Randomized Controlled Trial
Brief Title: Patient Activation Through Counseling, Exercise and Mobilization
Acronym: PACE-Mobil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Marta Kramer Mikkelsen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PACE-Mobil-PBL
Record Dates: First submitted 2018-01-10; First posted 2018-01-26 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Pancreas Cancer; Biliary Tract Cancer; Non Small Cell Lung Cancer; Advanced Cancer
Keywords: Older; Advanced Cancer; Exercise; Resistance training; Counseling; Mobilization
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to the intervention group and control group.
Who Masked: Outcomes Assessor
Masking Description: All physical tests will be conducted by masked health care professionals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (n=50) (Experimental): Participants in the intervention group will receive usual care and the multimodal and exercise-based intervention.
  Interventions: Behavioral: Multimodal and exercise-based intervention
- Control group (n=50) (No Intervention): Participants in the control group will receive usual care.

INTERVENTIONS:
Behavioral: Multimodal and exercise-based intervention — The multimodal and exercise-based intervention is comprised of:
  1. Supervised and group-based exercise two times a week (60 minutes per session). The program consists of warm-up, exercises for balance and flexibility, progressive resistance training, and stretching and relaxation.
  2. Individualized activity program based on step counts (with activity tracker). Based on each participant's starting point, preferences and motivation, an individualized program will be composed. Evaluation and goal-setting will be conducted once weekly.
  3. Nurse-led supportive and motivational counseling; each participant will be invited to two sessions of counseling (in week 1 + 6). Each session will be based on a holistic assessment of each participant's life situation. Advice and counseling will be provided based on identified problems and needs.
  4. A nutritional supplement (protein bar or drink) will be served to participants immediately after the supervised exercise session.
  Arms: Intervention group (n=50)

SUMMARY:
PACE-Mobil-PBL is a prospective randomized controlled trial. The aim is to investigate the effect of a multimodal and exercise-based intervention among older patients with advanced pancreatic cancer, biliary tract cancer, or lung cancer during treatment with first-line palliative chemotherapy, immunotherapy or targeted therapy.

The hypotheses: That the multimodal intervention will increase or maintain physical function levels and strength, reduce symptoms and side-effects, improve quality of life, reduce treatment-related complications and hospital admissions, and reduce risk of cancer cachexia and sarcopenia.

ELIGIBILITY:
Inclusion Criteria, participants must:

* Be diagnosed with locally advanced or metastatic pancreatic cancer, OR locally advanced or metastatic biliary tract cancer, OR locally advanced or metastatic non-small cell lung cancer within 12 weeks.
* Have unresectable cancer.
* Be treated with first-line palliative chemotherapy, immunotherapy or targeted therapy at the Department of Oncology, Herlev and Gentofte Hospital.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Have the ability to speak and read Danish, and to provide a signed informed consent form.

Exclusion Criteria, patients with:

* Small-cell lung cancer.
* Any physical condition that hinder the execution of physical exercise training.
* Documented and uncontrolled brain metastases that hinder participation in an exercise-based trial, based on the referring oncologist's assessment.
* Dementia, psychotic disorders, or other cognitive diseases or conditions that hinder participation in a clinical exercise-based trial.
* Unstable medical disease or history of serious or concurrent illness; any Medical condition that might be aggravated by exercise training or that cannot be controlled, including, but not restricted to congestive heart failure (NYHA class II-IV), unstable angina pectoris, implantable cardioverter defibrillator, or myocardial infarction within 6 months, based on the referring oncologist's assessment.

In patients with bone metastases:

- A bone metastatic burden or location that poses a risk of injury in the performance of exercise training, as assessed by the referring oncologist.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Lower body strength measured with the 30-second chair stand test | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Number of stands a participant can complete in 30-seconds from a seated position with their arms crossed over the chest. The assessments will be conducted by a blinded physiotherapist

SECONDARY OUTCOMES:
Recruitment rate | Up to 2 years
  Number of participants included from eligible patients
Adherence to exercise sessions | Up to 12 weeks
  Number of exercise sessions attended out of planned sessions
Adherence to counseling sessions | Up to 12 weeks
  Number of counseling sessions attended out of planned sessions
Adverse events | Up to 12 weeks
  Cases of exercise-related injuries or events, including, but not restricted to musculoskeletal-related events, falls, fall-related injuries, bleedings, or cardiovascular events.
Physical performance measured with the 6-minute-walk-test | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  The distance (measured in meters) a participant is able to walk over a total of six minutes on a hard flat surface. The assessments will be conducted by a blinded physiotherapist
Physical performance measured with the 6-meter Gait Speed Test | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  The assessments will be conducted by a blinded physiotherapist
Upper-body strength measured with the Handgrip Strength Test | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Handgrip strength will be measured using a hand-held Jamar dynamometer. The assessments will be conducted by a blinded physiotherapist
Physical activity level | Change measures (baseline, and 12 weeks).
  Step Counts (measured with Garmin Vivofit 3 activity tracker).
Qualitative assessment of participants' experiences | After 12 weeks
  Qualitative individual semi-structured interviews with participants from the intervention group
Quality of life | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Measured with the EORTC Quality of Life questionnaire (EORTC QLQ-C30)
Symptoms of depression | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Measured with the patient questionnaire 'Hospital Anxiety and Depression Scale' (HADS)
Symptoms of anxiety | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Measured with the 'Hospital Anxiety and Depression Scale' (HADS) patient questionnaire
Symptom burden | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Measured with the 'M.D. Anderson Symptom Inventory' patient questionnaire
Number of participants with side-effects to oncological treatment assessed with the Common Toxicity Criteria for Adverse Events version 4 | Up to 6 months
  Data will be collected from medical charts
Body weight | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Weight will be measured using standard procedures (no shoes, light clothing) and will be reported in kilograms
Body mass index | Change measures (baseline, 6 weeks, 12 weeks, and 16 weeks)
  Reported in kg/m^2
Whole-body Lean body mass (LBM) | Change measures (baseline, and 12 weeks)
  Measured with Bioimpedance and DXA scans
Whole-body fat mass | Change measures (baseline, and 12 weeks)
  Measured with Bioimpedance and DXA scans
Whole-body bone mineral density | Change measures (baseline, and 12 weeks)
  Measured with DXA scans
Inflammation (inflammatory biomarkers: C-reactive protein, Interleukin 6, YKL-40) | Up to 6 months
  Data will be collected from medical charts
Number of hospital admissions | Up to 6 months
  Data will be collected from medical charts
Causes of hospitalizations | Up to 6 months
  Data will be collected from medical charts
Length of hospitalizations (days) | Up to 6 months
  Data will be collected from medical charts
Survival | Up to 2 years
  Data will be collected from medical charts

CONTACTS AND LOCATIONS:
Overall Officials: Marta Kramer Mikkelsen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Herlev and Gentofte Hospital, Department of Oncology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mikkelsen MK, Lund CM, Vinther A, Tolver A, Ragle AM, Johansen JS, Chen I, Engell-Noerregaard L, Larsen FO, Zerahn B, Nielsen DL, Jarden M. Engaging the older cancer patient; Patient Activation through Counseling, Exercise and Mobilization - Pancreatic, Biliary tract and Lung cancer (PACE-Mobil-PBL) - study protocol of a randomized controlled trial. BMC Cancer. 2018 Sep 27;18(1):934. doi: 10.1186/s12885-018-4835-2. PMID 30261853